CLINICAL TRIAL: NCT05628584
Title: The Impact of High or Low FODMAP Diets on Postprandial Glucose Response and Gut Microbiota in Individuals With Prediabetes Treated With Metformin: A Randomized Crossover Controlled-Feeding Trial
Brief Title: High FODMAP Diet With Metformin in preDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elaine Chow (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor-Investigator, Elaine Chow, Clinical Assistant Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FODMAPMet
Record Dates: First submitted 2022-11-08; First posted 2022-11-28 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2022-11

CONDITIONS: PreDiabetes; Impaired Glucose Tolerance
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance | interventions — Metformin; FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High FODMAP (Experimental)
  Interventions: Combination Product: High FODMAP diet with metformin
- LOW FODMAP (Placebo Comparator)
  Interventions: Combination Product: Low FODMAP diet with metformin

INTERVENTIONS:
Combination Product: High FODMAP diet with metformin — Controlled High FODMAP diet (15g/day) from day 1-10, metformin XR 1000mg daily day 6-10 for each treatment period
  Arms: High FODMAP
Combination Product: Low FODMAP diet with metformin — Controlled low FODMAP diet (3g/day) from day 1-10, metformin XR 1000mg daily day 6-10 for each treatment period
  Arms: LOW FODMAP

SUMMARY:
This is a prospective, double blinded, randomised cross over feeding trial examine high or low FODMAP diet in combination with metformin on postprandial glucose responses and gastrointestinal tolerability and gut microbiota profiles.

The trial will compare high or low FODMAP diet, each of 10 days duration in combination with 5 days metformin, separated by a washout period of at least 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Body mass index 18 to 40 kg/m 2
3. Prediabetes defined as impaired fasting PG 5.6-6.9 mmol/l and/or impaired glucose tolerance with 2-hour PG 7.8-11.1 mmol/l on 75g oral glucose tolerance test (OGTT) and/or HbA1c 5.7-6.4% at screening

Exclusion Criteria:

1. Currently pregnant, lactating, as demonstrated by a positive pregnancy test at screening or planning pregnancy
2. Known current diabetes
3. Current or previous use of glucose-lowering or weight loss drugs in 3 months prior to screening
4. Concurrent participation in other weight loss or lifestyle intervention programmes
5. Current use or recent exposure to any medication that in the opinion of the investigator could have an influence on the patient's ability to participate in this study or on the performance of the test device.
6. Recent intake of prebiotic/probiotic or antibiotic, immunosuppressants (within 8 weeks of randomisation)
7. Extensive skin changes/diseases that preclude wearing the FGM on normal skin at the proposed application sites (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis).
8. Known uncontrolled thyrotoxicosis
9. Known vitamin B deficiency
10. Known irritable bowel syndrome or gastrointestinal disorders
11. Estimated glomerular filtration rate (eGFR) <45 ml/min/1.73m2 at screening
12. Current use of steroids
13. Have a known allergy to medical-grade adhesives
14. Known current or recent alcohol or drug abuse
15. Hypersensitivity to metformin
16. Acute or chronic metabolic acidosis, including diabetic ketoacidosis, with or without coma within 3 months of randomisation
17. Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection.
18. An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner).
19. Participants who are on a vegetarian or vegan diet as their habitual diet at screening.
20. Participants with clinically significant food allergy to components of the study diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Differences in postprandial glycemia | 10 days
  incremental area under curve on continuous glucose monitoring post meal

SECONDARY OUTCOMES:
Glucose response to 75g oral glucose tolerance test | 10 days
  fasting and postchallenge plasma glucose
Insulin response to 75g oral glucose tolerance test | 10 days
  insulin levels
Change in alpha diversity of gut microbiota | 10 days
  Changes in alpha diversity in gut microbiota
Change in beta diversity of gut microbiota | 10 days
  Changes in beta diversity in gut microbiota
Body weight | 10 days
  Differences in body weight between arms
Gastrointestinal symptoms | 10 days
  Measured on visual analogue scale 1-10 for each item, higher score indicates worse symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chu NHS, Ling J, Poon EWM, Lee JYS, Song Q, Zuo Z, Muir J, Chan JCN, Chow E. Combining a diet rich in fermentable carbohydrates with metformin improves glycaemic control and reshapes the gut microbiota in people with prediabetes. Nat Metab. 2025 Aug;7(8):1614-1629. doi: 10.1038/s42255-025-01336-4. Epub 2025 Jul 31. PMID 40745466